CLINICAL TRIAL: NCT02796937
Title: An Open-Label, Multicenter Study to Evaluate the Long-term Safety of Weekly Intravenous Alpha1-Proteinase Inhibitor (Human), Modified Process 60 mg/kg in Subjects With Pulmonary Emphysema Due to Alpha1-Antitrypsin Deficiency
Brief Title: Long Term Safety of Alpha1-Proteinase Inhibitor in Subjects With Alpha1 Antitrypsin Deficiency
Acronym: SPARTA-OLE
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GTi1201-OLE
Record Dates: First submitted 2016-06-03; First posted 2016-06-13 (Estimated); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Pulmonary Emphysema in Alpha-1 Antitrypsin Deficiency
Keywords: Pulmonary Emphysema; Alpha-1 Antitrypsin Deficiency; AATD; Alpha-1 PI Deficiency; Alpha-1 Proteinase Inhibitor
MeSH Terms: conditions — Pulmonary Emphysema; alpha 1-Antitrypsin Deficiency | interventions — Mp alpha1 receptor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (1):
- Alpha-1 MP (Experimental): Alpha-1 MP 60 mg/kg/week for up to 104 weeks
  Interventions: Biological: Alpha-1 MP

INTERVENTIONS:
Biological: Alpha-1 MP — Alpha-1 MP 60 mg/kg/week for up to 104 weeks
  Other Names: Prolastin-C

SUMMARY:
This is a 2-year open-label, multicenter extension of the double-blind, placebo-controlled GTi1201 study. The purpose of this study is to obtain an additional 2 years of safety data for intravenously administered Alpha1-MP 60 mg/kg/week in subjects with alpha1-antitrypsin deficiency (AATD).

DETAILED DESCRIPTION:
This is a 2-year open-label extension of the double-blind, placebo-controlled GTi1201 study. The purpose of this study is to obtain an additional 2 years of safety data for intravenously administered Alpha-1 MP 60 mg/kg/week in subjects with AATD.

The study consists of a Screening Visit (the same visit as the End-of-Study Visit in the GTi1201 study for subjects who complete the GTi1201 study or is the same visit as the Early Discontinuation Visit for subjects meeting the early withdrawal criterion for forced expiratory volume in 1 second [FEV1] decline), a treatment period of 104 weeks (beginning immediately after screening [on the same day as the Screening Visit] but no sooner than 1 week after the last infusion of investigational product in the GTi1201 study), and an End-of-Study Visit.

Subjects meeting the entrance criteria of the extension study will begin receiving weekly intravenous (IV) infusions of Alpha-1 MP 60 mg/kg on the day of screening and will continue to receive weekly infusions for a total of 104 infusions.

Safety assessments will include adverse events, concomitant medications, complete physical examination (excluding breast and genitourinary examination), hematology, chemistry, urine cotinine, and pregnancy test. Efficacy assessments will include whole lung computed tomography density, quality-of-life assessment, carbon monoxide diffusing capacity, and pulmonary function tests. The occurrence of chronic obstructive pulmonary exacerbations, will also be evaluated as a safety and as an efficacy measurement.

ELIGIBILITY:
Inclusion Criteria:

* Has completed participation in Study GTi1201 (ie, completed Week 156 and Week 160/End-of-Study Visit) OR has experienced a decline in FEV1 at the annualized rate of ≥134.4 mL/year at or after the Week 104 Visit in GTi1201.
* Is willing and able to provide informed consent

Exclusion Criteria:

* Is unable to physically or mentally undergo a CT scan (eg, unable to fit inside the CT scanner, claustrophobic).
* Has severe concomitant disease including, but not limited to, congestive heart failure and liver cirrhosis.
* Has primary and/or secondary (metastatic disease) pulmonary malignancy or other current malignancy with <1 year predicted overall survival.
* Has a metal object (newly received since starting GTi1201) that might interfere with chest CT quality and quantification. Metal objects include, but are not limited to, cardiac pacemaker, defibrillator, metal prosthetic heart valve, metal projectile, metal weapon fragments, or metal shoulder prosthesis.
* Is a female who is pregnant, breastfeeding or, if of child-bearing potential, unwilling to practice a highly effective method of contraception (oral, injectable, or implanted hormonal methods of contraception; placement of an intrauterine device or intrauterine system; condom or occlusive cap with spermicidal foam/gel/film/cream/suppository; male sterilization; or abstinence) throughout the study.
* Has clinical signs and symptoms of viral infection requiring virus safety testing at the Week 160/End-of-Study Visit or Early Discontinuation Visit in Study GTi1201, and the virus safety test results are indicative of acute or chronic infection with hepatitis A virus (HAV), hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV), or parvovirus B19 (B19V). Note: If the virus safety test results are indicative of acute or chronic infection with HAV, HBV, HCV, HIV, or B19V, the subject will be considered a screen failure and must be withdrawn from the study.
* Has current evidence of smoking, which includes electronic/vapor cigarettes, or has a positive urine cotinine test at the Week 160/End-of- Study Visit in Study GTi1201 that is due to smoking.
* Has current evidence of chronic alcoholism or illicit drug abuse (addiction).
* Is currently participating in another investigational product (IP) study.
* Has a history of anaphylaxis or severe systemic response to any plasma- derived alpha1-PI preparation or other blood product(s).
* In the opinion of the investigator, is likely to have compliance problems with the protocol and the procedures of the protocol.
* Has any medical condition that the investigator feels might confound the results of the study or pose an additional risk to the subject during study participation.

Ages: 20 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | Week 1 through Week 108
  Monitoring of AEs
Serious AEs (SAEs) | Week 1 through Week 108
  Monitoring of SAEs
Discontinuations from the study due to AEs | Week 1 through Week 108
  Monitoring of discontinuations due to AEs

SECONDARY OUTCOMES:
Change from baseline in whole lung PD15 (15th percentile point) | Week 1 through Week 104
  Whole lung PD15 measured by computed tomography scans
Change from baseline in carbon monoxide diffusing capacity (DLco) | Week 52 and Week 104
  DLco performed according to American Thoracic Society/European Respiratory Society (ATS/ERS) guidelines
Changes from baseline in forced expiratory volume in 1 second (FEV1) | Week 52 and Week 104
  FEV1 performed according to ATS/ERS guidelines
Change from baseline in Saint George's Respiratory Questionnaire | Week 52 and Week 104
  Health-related quality of life assessment tool
Incidence and severity of Chronic Obstructive Pulmonary Disease (COPD)exacerbations | Week 2 through Week 108
  Severe COPD exacerbations as defined by ATS/ERS guidelines
Change from baseline in the EQ-5D-5L Questionnaire | Week 52 and Week 104
  Heath-related quality of life assessment tool

CONTACTS AND LOCATIONS:
Locations (27):
- United States (6):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - University Of Miami Hospital, Doctors Office West Building, Miami, Florida
  - Accellacare, Wilmington, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Health Center at Tyler, Tyler, Texas
- Australia (5):
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Royal Adelaide Hospital, Adelaide
  - The Prince Charles Hospital, Chermside
  - St Vincent's Hospital Melbourne, Fitzroy
  - Institute for Respiratory Health Inc, Nedlands
- Canada (2):
  - Queen Elizabeth II Health Sciences Centre, Halifax
  - Inspiration Research Limited, Toronto
- Denmark (2):
  - Arhus Universitetshospital, Arhus C
  - Gentofte Hospital, Hellerup
- North Estonia Medical Centre Foundation, Tallinn, Estonia
- Turun yliopistollinen keskussairaala, Turku, Finland
- CHU Lyon - Hôpital Cardio-Vasculaire et Pneumologique Louis Pradel, Bron, Rhone, France
- New Zealand (3):
  - NZ Respiratory and Sleep Institute, Auckland
  - Christchurch Hospital NZ, Christchurch
  - Waikato Hospital, Hamilton
- Poland (2):
  - SPZOZ Szpital Uniwersytecki w Krakowie, Krakow
  - Instytut Gruzlicy i Chorob Pluc w Warszawie, Warsaw
- SBEI HPE Altai State Medical University of MoH and SD, Barnaul, Russia
- Sweden (3):
  - Sahlgrenska Sjukhuset, Gothenburg
  - Skånes Universitetssjukhus, Malmö, Malmo
  - Karolinska Trial Allicance, KTA Prim, Stockholm

IPD SHARING:
Plan to Share IPD: No